CLINICAL TRIAL: NCT00254670
Title: Naltrexone Effects on Alcohol Intake Using a Laboratory Bar in Asp40 Positive and Negative Alcohol Users Characterized by fMRI and Genetic Screening
Brief Title: Naltrexone Effects on Alcohol Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H5612-26059; H5612-26059
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2011-03

CONDITIONS: Social Drinker
Keywords: Alcohol; Naltrexone
MeSH Terms: interventions — Naltrexone

INTERVENTIONS:
Drug: Naltrexone

SUMMARY:
The purpose of this study is to examine drinking behavior and decision-making while taking Naltrexone and placebo. This is a double-blind, randomized, placebo-controlled crossover study. There are two cycles: one cycle on Naltrexone and one cycle on placebo.

DETAILED DESCRIPTION:
The study proposed is a 22 to 23 day, double-blind, placebo-controlled crossover study in 60 male and female moderate to heavy alcohol users who are Asp40 positive and negative. Subjects will undergo a 6 to 7-day cycle taking the first study drug (naltrexone or placebo) with an alcohol self-administration visit in the laboratory bar on the 6th or 7th day of drug. The first alcohol self-administration visit is followed by an 8 to 9 day washout period. Subjects then cross over to repeat the cycle while taking the other drug (placebo or naltrexone). On the final day (either day 8 or 9) of the first study drug cycle, the subject will undergo functional imaging (fMRI) at the WBIC. There will be at least one day in between the 'lab bar' and the fMRI scan. The first fMRI visit is followed by a 5-6 day washout period. Subjects then cross over to repeat the cycle while taking the other drug (placebo or naltrexone). Subjects will keep daily diaries of alcohol and medication use throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who are 21-40 years of age
* If female, 7-20 alcoholic drinks must be consumed weekly.
* If male, 10-25 alcoholic drinks must be consumed weekly.
* If female, must be non-lactating, not pregnant, and using a reliable contraception method (i.e. abstinence, intrauterine device [IUD], hormonal birth control, or double barrier method [male condom, female condom, or diaphragm plus a spermicidal agent such as contraceptive foam, jelly or cream]).
* Must have a body mass index (BMI) ≥18 and ≤30.
* Able and willing to provide an informed consent.
* Able to understand and follow the instructions of the investigator, including the delayed discounting tasks.
* Have a breath alcohol concentration of less than 0.02 on visits 1, 2, 3, 5, and 6; and 0.00 on visits 4, 4a, 7 and 7a.

Exclusion Criteria:

* Positive urine drug screen
* Using Cocaine, stimulants (other than nicotine and caffeine), methamphetamine, and/or amphetamines greater than 30 times in the last 24 months
* Using inhalants, hallucinogens, ecstasy, and/or ketamine greater than 30 times in the last 24 months
* Current enrollment in an alcohol, or other drug treatment program or current legal problems relating to alcohol, or other drug use, including awaiting trial or supervision by a parole or probation officer
* Binge drinking more than three times per week (>5 standard drinks in one session is a binge)
* Currently trying to quit alcohol use
* Current dependence on any other psychoactive drug (except nicotine or caffeine) and/or alcohol as determined by the study physician's assessment .
* Clinically significant medical or psychiatric illness as determined by screening blood tests, medical history, and physical exam performed by the study physician

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Primary Completion 2005-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Rowbotham, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States